CLINICAL TRIAL: NCT04605068
Title: Transverse Preputial Island Flap Versus Double Faced Preputial Flap for Repair of Penoscrotal Hypospadias With Chordee: A Randomized Controlled Trial
Brief Title: Transverse Preputial Island Flap Versus Double Faced Preputial Flap for Repair of Penoscrotal Hypospadias With Chordee
Acronym: DuckettvDFPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Al-Azhar Duckett's versus DFPF
Record Dates: First submitted 2020-10-09; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Hypospadias, Penoscrotal; Chordee
Keywords: Penoscrotal Hypospadias; Chordee; Tubularized Double-Faced Preputial Flap; Duckett's Urethroplasty; One-Stage Repair
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Intervention Model Description: 144 patients will be randomly divided (using the computer-generated randomization table) into two equal groups, each will include 72 patients; Group I will undergo transverse preputial island flap (Duckett's technique) and Group II will undergo double-faced preputial flap (DFPF).
Who Masked: Participant, Investigator
Masking Description: Double masking (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverse preputial island flap (Duckett's technique) (Active Comparator): 72 patients (Group I) with penoscrotal hypospadias with chordee
  Interventions: Procedure: Transverse preputial island flap (Duckett's technique)
- Double-faced preputial flap (DFPF) (Active Comparator): 72 patients (Group II) with penoscrotal hypospadias with chordee
  Interventions: Procedure: Double-faced preputial flap (DFPF)

INTERVENTIONS:
Procedure: Transverse preputial island flap (Duckett's technique)
  Arms: Transverse preputial island flap (Duckett's technique)
Procedure: Double-faced preputial flap (DFPF)
  Arms: Double-faced preputial flap (DFPF)

SUMMARY:
The purpose of this study is to compare the outcomes and complications of the transverse preputial island flap (Duckett's procedure) to those of double-faced preputial flap (DFPF) for one-stage repair of penoscrotal hypospadias with chordee, in addition to clinical functional evaluation by estimated urine flow.

DETAILED DESCRIPTION:
Type of study: RCT

Review of literature:

* Different modalities of urethroplasty for repair of proximal hypospadias with chordee (two-stage repair, one-stage repair, flap, graft).
* Disadvantages of two-stage urethroplasty for proximal hypospadias with chordee..
* Merits of one-stage urethroplasty for proximal hypospadias with chordee. This is a prospective randomized controlled study conducted at pediatric surgery department, Al-Houssain & New Damietta Al-Azhar University Hospitals, from March 2014 to March 2020, on 144 male patients with penoscrotal hypospadias with chordee. Patients will be investigated by routine laboratory tests for fitness for surgery. All of them will undergo one-stage repair using either of 2 techniques of tubularized preputial flap; Duckett's versus DFPF. Written informed consent will be obtained from parents of all participants in the study.

Institutes of the study:

A multicenter study at Pediatric Surgery Departments, Al-Azhar University hospitals in Cairo and New Damietta. Number of cases: One-hundred-Forty four male patients. Time frame: period of 6 years.

Ethical Consideration:

The protocol will be discussed and approved for clinical study by the Ethical Research Committee at the principal investigator's hospital. The procedures and the aim of the study will be clearly explained to the patient and the family. A written informed consent will be obtained before enrollment of the patients into the study. The family refusal to give consent for one-stage repair is respected but does not deprive the patient from getting surgical care by two-stage repair.

Preoperative preparation:

All patients will be subjected to history taking, clinical examination, and necessary laboratory investigations (CBC, Coagulation profile, Liver and Renal Function tests, Electrolytes Panel, Urinalysis). They will receive a dose of single broad-spectrum antibiotic 30 min-1 hour before surgery. Patients will be randomly divided (using the computer-generated randomization table) into two equal groups, each will include 72 patients; Group I will undergo transverse preputial island flap (Duckett's technique) and Group II will undergo double-faced preputial flap (DFPF). Both techniques will be done by all members of the surgical team equally.

Follow-up:

Patients will be followed-up at OPD.

Statistical Analysis:

Data were collected using a data collecting sheets (annexes) and were analyzed using the statistical package for social sciences (SPSS) version 24.0 (IBM SPSS Statistics for Windows, IBM Corp, Armonk, NY, USA). Continuous variables were expressed as mean±standard deviation (SD), range, and average and categorical variables were expressed as frequency count & percentage. Fisher's exact test was used for comparison of frequency counts/percentage. A two-sided p-value < 0.05 was considered statistically significant.

Discussion:

It will focus on one-stage urethroplasty using the preputial flap for proximal hypospadias with chordee. The results obtained from this study will be compared between both group and with those reported in the literature.

Also, it will focus on results, complications, their management, and clinical evaluation by estimated urine caliber and micturition time. At the end, the investigators will conclude the reconstructive technique that gives the better results and least morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Uncircumcised male patients with penoscrotal hypospadias,
* rudimentary urethral plate
* with moderate-to-severe chordee and
* no history of previous repair

Exclusion Criteria:

* circumcised patients,
* patients with other types of hypospadias such as glanular or distal shaft or
* with mild chordee corrected after penile degloving,
* recurrent hypospadias, or
* lost to follow-up.

Ages: 6 Months to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male children with penoscrotal hypospadias with chordee
Enrollment: 144 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Urethrocutaneous fistula (number & percent) | 2 years
  Urethrocutaneous fistula
Meatal stenosis (number & percent) | 2 years
  Meatal stenosis
Urethral stricture (number & percent) | 3 years
  Urethral stricture

SECONDARY OUTCOMES:
Penile rotation (number & percent) | 3 years
  Penile rotation
Urine stream (in caliber) | 3 years
  Urine stream
Urine stream (in meters) | 3 years
  Urine stream
Micturition time (in seconds) | 3 years
  Micturition time
Follow-up period (in months) | 5 years
  Follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Shahin, MD, Principal Investigator — Al-Azhar New Damietta University

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for other researchers including methodology, figures, tables, results, and philosophy of discussion and the value this study will add to the literature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: March 2020 till indefinitely
Access Criteria: after the article became accepted and available online.